CLINICAL TRIAL: NCT06111508
Title: An Exploratory 16-Week Pilot Study of the Effect and Safety of a Novel CGM-Based Titration Algorithm for Basal Insulin, With or Without Non-Insulin Antidiabetic Drugs, in Type 2 Diabetes Mellitus Participants Treated With Basal Insulin.
Brief Title: The Effect and Safety of a Novel CGM-Based Titration Algorithm for Basal Insulin in T2DM Participants.
Acronym: CGM-DTx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Marc Breton, Principal Investigator, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 230357
Record Dates: First submitted 2023-10-26; First posted 2023-11-01 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes; Continuous Glucose Monitoring (CGM); Degludec Insulin; Self-monitoring blood glucose (SMBG)
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Intervention Model Description: Multi-center, randomized, parallel group, active-comparator clinical trial of CGM based titration of insulin Degludec vs. standard titration by SMBG.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Continuous Glucose Monitoring (CGM) based Titration (Experimental): The CGM-based titration algorithm will run on the Diabetes Assistant and Amazon Web Services (AWS) platform (DiAs-Cloud). DiAs-Cloud enables the seamless integration of a smart phone application and AWS server architecture to enable data capture, dose computation, review by the clinical team, and communication to study participants. For dose computation the algorithm is comprised of three components; titration glucose level, personalized target, and safety hypoglycemia feature.
  Interventions: Device: Continuous Glucose Monitoring (CGM)-based titration algorithm implemented in DiAs
- Standard Self-Monitoring Blood Glucose (SMBG) Titration (No Intervention): The SMBG-based titration algorithm will run on the Diabetes Assistant and Amazon Web Services (AWS) platform (DiAs-Cloud). DiAs-Cloud enables the seamless integration of a smart phone application and AWS server architecture to enable data capture, dose computation, review by the clinical team, and communication to study participants. Participants in the standard SMBG based titration group will wear a blinded CGM during the whole study. The total daily basal insulin dose will be converted 1:1 to Degludec. Algorithm informed dose changes will be made once weekly and checked by study physician.

INTERVENTIONS:
Device: Continuous Glucose Monitoring (CGM)-based titration algorithm implemented in DiAs — A Continuous Glucose Monitoring (CGM)-based once weekly titration algorithm of basal insulin as implemented in DiAs Cloud platform
  Other Names: Degludec
  Arms: Continuous Glucose Monitoring (CGM) based Titration

SUMMARY:
The goal of this clinical trial is to compare the effect of a continuous glucose monitor (CGM) based titration algorithm to standard titration by self-monitoring blood glucose (SMBG) in participants with Type 2 Diabetes already using long acting insulin. The comparison aims to study the difference in glycemic control between the two therapies. Participants will be followed for 18 weeks and will be provided with Degludec insulin, insulin pen, and a CGM (Dexcom G6).

DETAILED DESCRIPTION:
This is an 18-week study designed to investigate the effect of a continuous glucose monitor (CGM) based titration algorithm versus a standard titration by self-monitoring blood glucose (SMBG) on glycemic control in Type 2 Diabetes (T2DM) participants using insulin Degludec. After 2 weeks of blinded CGM baseline observation, participants are randomized 2:1 to CGM-based titration or standard titration by SMBG for 16 weeks. In the SMBG group, all titrated doses will be reviewed by a study physician prior to use and participants will wear a blinded CGM during the whole study. After completion of the 16-week titration, participants are followed up for 2 days. Participants will be divided related to use of sulfonylureas or glinides with a maximum cap of nine participants being treated with sulfonylureas and glinides to complete the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older at signing of informed consent
2. Diagnosis of Type 2 Diabetes minimum 180 days before the day of screening
3. Hemoglobin A1c between 7-9% and measured by local lab at screening
4. On daily basal insulin for at least 90 days before inclusion into the study
5. Stable dose of oral and injectable (other than insulin) antidiabetic medications for 90 days prior inclusion. Acceptable medications include:

   1. Metformin
   2. Sulfonylureas
   3. Meglitinides (glinides)
   4. Dipeptidyl peptidase 4 (DPP-4) inhibitors
   5. Sodium glucose co-transporter 2 (SGLT2) inhibitors
   6. Thiazolidinediones
   7. Alpha-glucosidase inhibitors
   8. Oral combination products (for the allowed individual oral anti-diabetic drugs)
   9. Oral or injectable Glucagon-like peptide-1 (GLP-1) Receptor Agonists (RAs)
   10. If on sulfonylureas or glinides, willingness to reduce dose by 50%

Exclusion Criteria

1. Hypersensitivity to Degludec
2. Use of an insulin pump
3. Use of a short-acting insulin
4. Participation or has participated in another trial within 90 days of the screening visit
5. Female who is pregnant or intends to become pregnant or is of child-bearing potential and not using an adequate contraceptive method
6. Any disorder, except for conditions associated with T2D, which in the investigator's opinion might jeopardize participant's safety or compliance with the protocol.
7. Treatment with any medication for the indication of diabetes or obesity other than stated in the inclusion criteria within 90 days of the screening visit
8. Known skin reactions to CGM adhesives
9. Current/prior use of CGM within 30 days of the screening visit
10. Any planned surgery or procedures where basal insulin would be decreased or held in anticipation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-11-29 (Actual); Primary Completion 2024-09-13 (Actual); Study Completion 2024-09-16 (Actual)

PRIMARY OUTCOMES:
Change in Time in Range | From baseline (-2 to 0 weeks) to weeks 14-16 (2 weeks)
  Change in CGM-measured time in range 3.9-10.0 mmol/L (70-180 mg/dL) from baseline to weeks 14-16, compared between control and experimental arm.

SECONDARY OUTCOMES:
Change in HbA1c | From week 0 to week 16
  Percent change in HbA1c
Change in Time in Tight Range | From baseline (week -2-0) to week 14-16
  Percent change in time in tight range 3.9-7.8 mmol/L (70-140 mg/dL)
Change in Time above 10.0 mmol/L (180 mg/dL) | From baseline (week -2-0) to week 14-16
  Percent of time spent above 10.0 mmol/L (180 mg/dL).
Change in Time above 13.9 mmol/L (250 mg/dL) | From baseline (week -2-0) to week 14-16
  Percent of time spent above 13.9 mmol/L (250 mg/dL)
Change in Continuous Glucose Monitoring Coefficient of variation (%) | From baseline (week -2-0) to week 14-16
  The statistical measure (%) of the relative dispersion of data points in a data series around the average CGM-measured blood glucose level.
Change in Mean Glucose Level | From baseline (week -2-0) to week 14-16
  The average CGM-measured blood glucose level (mmol/L).
Change in Time below 3.9 mmol/L (70 mg/dL) | From baseline (week -2-0) to week 14-16
  Percent of time spent below 3.9 mmol/L (70 mg/dL).
Change in Time below 3.0 mmol/L (54 mg/dL) | From baseline (week -2-0) to week 14-16
  Percent of time spent below 3.0 mmol/L (54 mg/dL).
Frequency of Hypoglycemic Events | From week 0 to week 16
  The number of clinically significant hypoglycemic episodes (level 2) (<3.0 mmol/L (54 mg/dL), confirmed by BG meter) or severe hypoglycemic episodes (level 3).
Frequency of Serious Adverse Events | From week 0 to week 16
  The number of serious adverse events (SAEs).
Frequency of Treatment Emergent Adverse Events | From week 0 to week 16
  The number of treatment emergent adverse events (TAEs).
Frequency of Device Deficiencies | From week 0 to week 16
  The number of device deficiencies (DDs). A device malfunction is any failure of a device to meet its performance specifications or otherwise work as intended. Performance specifications include all claims made in the labelling for the device. The intended performance of a device refers to the intended use for which the device is labelled or marketed.
Percent Acceptance Rate | From week 0 to week 16
  Investigator acceptance rate of weekly dose guidance - from CGM-based titration (Experimental arm only).
Frequency of Dose Changes | From week 0 to week 16
  The investigator changes the dose from the recommended or the current dose (Experimental arm only).

CONTACTS AND LOCATIONS:
Overall Officials: Ralf M Nass, MD, Study Chair — University of Virginia
Locations (2):
- United States (2):
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Will follow the NIH Data Sharing Policy and Implementation Guidance on sharing research resources for research purposes to qualified individuals in the scientific community.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available after the primary publications of each study.
Access Criteria: The Data Sharing Agreements will be formulated by the study team.

REFERENCES:
- [Derived] El Fathi A, Nass R, Levy CJ, Levister C, O'Malley G, Shah NA, Hassan S, Quainoo C, Koravi CLK, Nguyen TN, Santini GM, Emory E, Alix C, Flanagan DK, Fulkerson D, Clancy Oliveri M, Laugesen C, Lindelov JK, Hansen PW, Breton MD. Safety and Feasibility of Algorithmic Continuous Glucose Monitoring-Based Titration in People with Type 2 Diabetes Using Insulin Degludec, With or Without Noninsulin Glucose-Lowering Drugs: A 16-Week Randomized Controlled Trial. Diabetes Technol Ther. 2026 Feb 6:15209156261420193. doi: 10.1177/15209156261420193. Online ahead of print. PMID 41651803

DOCUMENTS (1):
  • Informed Consent Form (2024-02-19): https://cdn.clinicaltrials.gov/large-docs/08/NCT06111508/ICF_000.pdf